CLINICAL TRIAL: NCT04469608
Title: Establishing TCM Daycare Model and Teaching Mechanism of Depression Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH109-REC3-041
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Traditional Chinese Medicine; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Acupuncture Therapy; Yoga; Mindfulness; Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM clinical daycare model for depression patients (Experimental): Tai Chi and Acupuncture and Yoga and Mindfulness
  Interventions: Behavioral: acupuncture
- Depression patients (No Intervention): Tai Chi and acupuncture and yoga and mindfulness are not added

INTERVENTIONS:
Behavioral: acupuncture — Traditional Chinese medicine clinical daycare
  Other Names: yoga; mindfulness; Tai Chi
  Arms: TCM clinical daycare model for depression patients

SUMMARY:
The teaching platform of the TCM daycare clinics for depression patients will provide a good clinical training environment for the trainees. They can learn how to take care of depression patients by the lectures and the clinical practice experiences in the daycare clinics. They can also learn a holistic approach, a patient-centered healthcare service. This teaching model will strengthen the clinical training of TCM and enhance the international competitiveness of TCM doctors.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a serious psychiatric illness with a high lifetime prevalence rate and causes major clinical, social and economic burden to patients and their family. Despite that more than 40 antidepressants with various mechanisms are available on the market, half of patients fail to achieve remission with optimized medication treatment because of unsatisfactory efficacy, frequent intolerability and poor compliance of pharmacotherapies. However, Traditional Chinese medicine (TCM) is a safe and effective therapy which has many previous evidences to improve the treatment of depression. The aim of this project is to build up a TCM clinical daycare model for depression patients, and to establish a teaching platform for TCM trainees.

The TCM daycare model will be provided by a team organized by doctors, nurses, pharmacists, psychologist, nutritionist and case managers. This model will provide a comprehensive TCM care system to improve the clinical symptoms and quality of life of depression patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of depression according to DSM-IV (Diagnosis code: 296.21-296.30, 300.4)
2. Age 18-65 years, male or female
3. Evaluation of the 21-item Hamilton Rating Scale for Depression (HAMD) 8 points or more
4. Fully understand the entire research plan and sign the informed consent form (aged 18-20 years old must be jointly signed by a legal agent)

Exclusion Criteria:

1. Have a diagnosis of mental illness other than depression in the last or past 6 months, including unipolar major depression, including dyslexia, organic mental disorder, impulse control disorder, substance use disorder, bipolar mental disorder or substance abuse.
2. Medical history of patients diagnosed with borderline, antisocial personality disorder
3. Take anti-psychotic disorders and anti-epileptic drugs in the past six months.
4. Have or may become pregnant
5. A person with serious suicidal ideation or suicide attempt who must be hospitalized for close monitoring

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale, HAM-D | Start of treatment (day 0) and end of treatment (week 8)
  Each question of HAM-D is rated 3-5 points, eight questions are 0-2 points, nine questions are 0-4 points, and the total score is 0-52 points. Evaluate the emotional and physical and mental states observed in the case during the most recent week and interview.
Beck Depression Inventory(BDI) | Start of treatment (day 0) and end of treatment (week 8)
  Beck Depression Inventory assesses the degree of depression of 13-80 year olds, as a diagnosis and treatment reference
Pittsburgh Sleep Quality Inventory | Start of treatment (day 0) and end of treatment (week 8)
  It is suitable for the evaluation of sleep quality in patients with sleep disorders and mental disorders, and is also suitable for the evaluation of sleep quality in ordinary people.
WHOQOL-Taiwan | Start of treatment (day 0) and end of treatment (week 8)
  Four-dimension: Physiology + Independence; Psychology + Spirituality/Religion/Personal Belief;

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Lee, Study Director — Department of Acupuncture, China Medical University Hospital Taichung, Taiwan
Locations (1):
- Department of Acupuncture, China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No